CLINICAL TRIAL: NCT01913678
Title: The Effect of Dairy Fat and Inulin on Fasting Induced Adipose Factor (FIAF) Blood Concentrations
Acronym: FIAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Arla Foods (Industry)
Responsible Party: Principal Investigator, Arne Astrup, Prof., MD, Head of Department, Department of Nutrition, Exercise and Sports, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B307
Record Dates: First submitted 2013-07-30; First posted 2013-08-01 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Inulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Inulin (Active Comparator): The participants will be given all dietary items in their diet. In the inulin arm, approximately 15 grams of inulin will be included in the diet.
  Interventions: Other: Inulin; Other: Complete diet
- Whole milk (Active Comparator): The participants will be given all dietary items in their diet. In the whole milk arm, approximately 1 liter of whole milk will be included in the diet.
  Interventions: Other: Complete diet; Other: Whole milk
- Complete diet (Placebo Comparator): The participants will be given all dietary items in their diet.
  Interventions: Other: Complete diet

INTERVENTIONS:
Other: Inulin — The participants will be given all dietary items in their diet. In the inulin arm, approximately 15 grams of inulin will be included in the diet.
  Arms: Inulin
Other: Complete diet — The participants will be given all dietary items in their diet with no additional products.
Other: Whole milk — The participants will be given all dietary items in their diet. In the whole milk arm, approximately 1 liter of whole milk will be included in the diet.
  Arms: Whole milk

SUMMARY:
The objective of this study is to investigate whether intake of a diet with a high content of butyrate (from dairy fat) can affect blood FIAF concentration compared to a control diet. Further to examine whether high intake of inulin (a prebiotic) can increase the proportion of butyrate-producing bacteria in the gut and thereby affect blood FIAF concentration. In addition, the correlation between FIAF blood concentrations and resting energy expenditure, blood lipid profile and gut microbiota composition will be investigated.

Furthermore, this study will investigate whether the source of FIAF can be determined. To this end, adipose tissue biopsies will be analyzed and an in vitro experiment with fecal water samples will be carried out.

The study is a crossover randomized controlled trials with 3 arms. Each arm has a duration of 3 weeks. 20 overweight/obese subjects will be enrolled into the study and randomized to the order of interventions. Before and after each intervention period, blood samples will be collected and the participants will have their resting metabolic rate measured. At the end of each intervention period, the participants will collect feces for 5 consecutive days. In addition, adipose tissue biopsies will be taken after each intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Age: 23-45
* BMI: 25-32 kg/m2
* Body fat percentage (BFP) > 25

Exclusion Criteria:

* Chronic diseases (known diabetes, cardiovascular disease (CVD), Intestinal Bowel Disease and other chronic diseases likely to affect the results of the present study)
* Milk allergy/lactose intolerance
* Intolerance towards inulin
* Fasting glucose ≥7.0 mmol/l or non-fasting glucose ≥ 11 mmol/l*
* Use of antibiotics 2 months before commencement of study
* Use of dietary supplements incl. multivitamins during run-in and the entire study period
* Smoking
* Elite athletes (>10 hours of strenuous physical activity per week)
* Use of prescription medicine which could affect the results of the present study, including systemic glucocorticoids
* Use of lipid-lowering agents or medication with contraindications for a high fat diet
* Blood pressure > 140/90 mmHg
* Blood donation <1 month before study commencement and during study period
* Simultaneous participation in other clinical studies
* Inability, physically or mentally, to comply with the procedures required by the study protocol, as evaluated by the study staff

Ages: 23 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07-03 (Actual); Study Completion 2014-07-03 (Actual)

PRIMARY OUTCOMES:
Changes in FIAF blood concentration | 21 days

SECONDARY OUTCOMES:
Changes in blood lipid profile including triglyceride, free fatty acid, low density lipoprotein cholesterol (LDL-C), high density lipoprotein cholesterol (HDL-C), glycerol, butyrate | 21 days
Changes in microbiotic composition and characterization of gut microbiota, including metabolites | 21 days
Changes in short-chain fatty acid content of feces (butyrate, propionate and acetate) | 21 days
Changes in resting energy expenditure/lipid oxidation | 21 days
Changes in parameters involved in glucose metabolism | 21 days
Changes in FIAF adipose tissue messenger ribonucleic acid (mRNA) levels | 21 days
Changes in gene expression and protein concentration of genes/proteins related to obesity, lipid metabolism, adipocyte differentiation, hypoxia and FIAF signaling in adipose tissue | 21 days
Changes in FIAF mRNA/protein expressed in or secreted from human intestinal cell lines | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, Prof., MD, Principal Investigator — Department of Nutrition, Exercise and Sports
Locations (1):
- Department of Nutrition, Exercise and Sports, Frederiksberg, Copenhagen, Denmark

REFERENCES:
- See also: Related Info — http://sfx.aub.aau.dk/sfxaub?sid=google&auinit=T&aulast=Bl%C3%A6del&atitle=A+randomised,+controlled,+crossover+study+of+the+effect+of+diet+on+angiopoietin-like+protein+4+(ANGPTL4)+through+modification+of+the+gut+microbiome&id=doi:10.1017/jns.2016.38